CLINICAL TRIAL: NCT00005229
Title: HIV-Associated Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1109; R01HL041507 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Diseases; Acquired Immunodeficiency Syndrome; HIV Infections
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Cardiomyopathies; Acquired Immunodeficiency Syndrome; HIV Infections

SUMMARY:
To develop natural history data regarding the incidence, clinical course, prognosis, and effects of treatment with anti-viral and immunosuppressive agents on HIV-associated heart disease. A second part of the study evaluated a number of possible mechanisms underlying the development of HIV heart disease.

DETAILED DESCRIPTION:
BACKGROUND:

As AIDS reached epidemic proportions it became apparent that heart disease contributed to morbidity in this disease. By 1988, survival following diagnosis with AIDS had improved, and the impact of heart disease on quality of life and survival in these patients had increased in parallel. The spectrum of pathology which comprised AIDS heart disease was diverse and the contribution of cardiac disease to mortality was quite unclear. Unanswered questions included: which seropositive individuals would develop heart disease; what was the spectrum of heart disease in these patients; were there any useful parameters for risk stratification; what was the clinical course; was the etiology due to HIV or other infectious agents or immunologic; did anti-viral agents or immunosuppressive treatment affect the disease course?

This project was part of an Institute-initiated study on AIDS-Associated Heart Disease in Adults. The concept was approved by the National Heart, Lung, and Blood Advisory Council in September 1987. The Request for Applications was also released in September 1987. Awards were made in July 1988.

DESIGN NARRATIVE:

Asymptomatic patients were recruited from the azidothymidine (AZT) versus placebo trial, open label AZT trial, isoprinosine versus placebo trial, and Ampligen versus placebo trial at George Washington University Medical Center. Symptomatic patients were referred from nearby clinics. Baseline information collected included age, sex, weight, HIV risk factors, dates of seroconversion, total CD4 lymphocyte count, clinical symptoms, symptoms of AIDS-related complex, first opportunistic infection, development of tumors or neurologic symptoms, anti-viral therapy, chest pain, symptoms of and treatment for congestive heart failure, evidence of arrhythmia, and initiation of anti-arrhythmic therapy. Date and cause of death were recorded along with autopsy findings. Non-invasive serial electrocardiograms and echocardiograms were performed in all participants at baseline and every four months. Endomyocardial biopsy was performed in patients with congestive cardiomyopathy, those with echocardiographic evidence of left ventricular dysfunction or large pericardial effusions, and those with significant arrhythmias. Endomyocardial biopsies were obtained from ten asymptomatic individuals, five of whom had lymphadenopathy, and five of whom had no lymphadenopathy. Percutaneous pericardiocentesis was performed in patients with large pericardial effusions to obtain samples for bacterial, mycobacterial, HIV and cytomegalovirus cultures. The fact that the majority of these patients were participating in clinical trials of various anti-viral agents allowed evaluation of their effects on the development of heart disease. The second part of the project was a study of the pathogenesis of HIV-associated heart disease. Light and electron microscopic findings were examined in the heart at various clinical stages of HIV infection. Cardiocytes were examined for presence of HIV and other infectious agents.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1988-07; Study Completion 1993-06 (Actual)

REFERENCES:
- [Background] Turco M, Seneff M, McGrath BJ, Hsia J. Cardiac tamponade in the acquired immunodeficiency syndrome. Am Heart J. 1990 Dec;120(6 Pt 1):1467-8. doi: 10.1016/0002-8703(90)90271-x. No abstract available. PMID 2248200
- [Background] Hsia J, Goldstein AL, Simon GL, Sztein M, Hayden FG. Peripheral blood mononuclear cell interleukin-2 and interferon-gamma production, cytotoxicity, and antigen-stimulated blastogenesis during experimental rhinovirus infection. J Infect Dis. 1990 Sep;162(3):591-7. doi: 10.1093/infdis/162.3.591. PMID 2167330
- [Background] Porter-Jordan K, Rosenberg EI, Keiser JF, Gross JD, Ross AM, Nasim S, Garrett CT. Nested polymerase chain reaction assay for the detection of cytomegalovirus overcomes false positives caused by contamination with fragmented DNA. J Med Virol. 1990 Feb;30(2):85-91. doi: 10.1002/jmv.1890300202. PMID 2156009
- [Background] Rodriguez ER, Nasim S, Hsia J, Sandin RL, Ferreira A, Hilliard BA, Ross AM, Garrett CT. Cardiac myocytes and dendritic cells harbor human immunodeficiency virus in infected patients with and without cardiac dysfunction: detection by multiplex, nested, polymerase chain reaction in individually microdissected cells from right ventricular endomyocardial biopsy tissue. Am J Cardiol. 1991 Dec 1;68(15):1511-20. doi: 10.1016/0002-9149(91)90288-v. PMID 1746436
- [Background] Hsia J, Colan SD, Adams S, Ross AM. Late potentials and their relation to ventricular function in human immunodeficiency virus infection. Am J Cardiol. 1991 Nov 1;68(11):1216-20. doi: 10.1016/0002-9149(91)90196-r. PMID 1951082
- [Background] Hsia J, Ross AM. Pericardial effusion and pericardiocentesis in human immunodeficiency virus infection. Am J Cardiol. 1994 Jul 1;74(1):94-6. doi: 10.1016/0002-9149(94)90501-0. No abstract available. PMID 8017317